CLINICAL TRIAL: NCT06096740
Title: The Effects of Trauma-focused Psychotherapy on Reward Circuitry Function and Information Encoding
Brief Title: Psychotherapy Effects on Reward Processing in PTSD
Acronym: PERPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Greg Fonzo, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00004746
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Post Traumatic Stress Disorder; Diminished Pleasure; Anhedonia; PTSD; Chronic PTSD; Chronic Post-Traumatic Stress Disorder
Keywords: PTSD; Post Traumatic Stress; Emotional Numbing; CPT; Cognitive Processing Therapy; Therapy; Chronic PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anhedonia | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified based upon baseline presence/absence of MDD and will occur using pre-specified block randomization with randomly-sized blocks of either 4 or 6 to ensure near-equal distribution of participants with and without comorbid MDD between the two arms over time, while avoiding the ability for study personnel to predict treatment assignment of the next participant. Blocks will involve various orderings of participant assignment, each block will be assigned a number, and a random list generator will then order the block sequences prior to the start of the study. This will ensure equal numbers of participants with and without MDD are assigned to each treatment condition and limit predictability of assignment.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: As participants will necessarily be aware of their arm assignment, symptom raters (research assistants) and study therapists will be blinded to participant arm assignment to reduce risk of ascertainment bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Those individuals randomized to immediate treatment will commence individual cognitive processing therapy (CPT) with an assigned study therapist, following the completion of baseline procedures.
  Interventions: Behavioral: Cognitive Processing Therapy
- Delayed Treatment (Placebo Comparator): Individuals randomized to the delayed treatment condition will be informed after randomization that their treatment will start in 6-8 weeks (the approximate period it will take for individuals in the immediate treatment arm to complete CPT and post-treatment assessments).
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive processing therapy is a widely-utilized, empirically-supported treatment developed for PTSD. It is based on a cognitive theory of trauma which emphasizes the impact of trauma on belief systems and the development of "stuck points", which are unhealthy, unrealistic, and maladaptive ways of thinking that serve to maintain unhealthy beliefs and reinforce PTSD symptoms.
  Other Names: CPT

SUMMARY:
The purpose of this study is to identify how trauma-focused psychotherapy changes the function of brain circuitry in posttraumatic stress disorder (PTSD) and how this mediates improvements in the diminished ability to experience positive emotions following a traumatic or extremely stressful life event. In this instance, the investigators will be using cognitive processing therapy (CPT), a widely-utilized and evidence-based treatment for PTSD.

DETAILED DESCRIPTION:
The goals of the study are as follows:

1. Quantify, under conditions of safety (no threat), how PTSD psychotherapy alters reward circuit function and information encoding.
2. Identify how presence of threat augments PTSD psychotherapy effects on reward circuit function and information encoding.
3. (Exploratory). Identify how, following psychotherapy, changes in reward circuit function and information encoding under conditions of safety and threat are associated with improvements in symptoms of diminished positive affect (DimPA).

To accomplish the goals of the study, the investigators propose a neuroimaging-coupled, randomized clinical trial of immediate vs. delayed individual cognitive processing therapy (CPT) in individuals (N=120) with a primary diagnosis of chronic PTSD. Individuals will undergo, prior to randomization, clinical and neurobiological assessment with functional magnetic resonance imaging (fMRI) during completion of several reward processing paradigms. Two of these involve both a normal "safe" context and a threat context manipulation (threat of mild electrodermal shock that is periodically cycled throughout the task). Another paradigm involves making decisions to either approach reward or forego a reward when this decision conflicts with the likelihood of an aversive outcome. This is known as approach-avoidance conflict (AAC). This battery will provide a comprehensive characterization of reward processing behavior and circuit function and establish its relationship to treatment processes, as well as how such processes may vary as a function of threat.

ELIGIBILITY:
Inclusion Criteria:

* English as primary language, and comprehension suitable to understand experimenter instructions.
* Current and chronic syndromic PTSD, defined as being exposed to a DSM-5 Criterion A traumatic event, with the presence DSM-5 qualifying PTSD symptoms for at least 3 months, as assessed by the Clinician-Administered PTSD Scale for DSM-5.
* Able and willing to undergo functional magnetic resonance imaging (fMRI).
* Willingness to participate in repeated assessments and as part of a delayed treatment group.

Exclusion Criteria:

* Evidence of current or prior history of psychosis or bipolar disorder as evidenced by self-report or clinical interview.
* Active substance dependence within the past 6 months as evidenced by clinical interview.
* Current regular psychiatric medication use (i.e. antidepressants), except for as-needed benzodiazepine or opiate medication no more than three times per week, on average, or for short-duration stimulant medication for attention deficit hyperactivity disorder that can be skipped within 24 hours of study visits.
* A recent (<6 months) suicide attempt or current active ideation with intent.
* Unremovable ferrous metal in body.
* History of neurological disorder, stroke, seizures/convulsions (except febrile seizures in childhood), epilepsy, brain surgery, electroconvulsive or radiation treatment, brain hemorrhage or tumor, or thyroid disorder.
* Anyone who is pregnant or trying to become pregnant.
* Current or past year (> 3 sessions), psychotherapy with a prominent exposure or cognitive restructuring component.
* Previous or current (es)ketamine treatment and/ or brain stimulation/neuromodulation treatment.
* Other ongoing treatment that is likely to confound experimental effects.
* Previous penetrating head injury/traumatic brain injury. Mild-to-moderate traumatic brain injury without penetrating injury is allowable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Within subject beta coefficients for each parametrically modulated regressor of the Reinforcement Learning Task with Threat | [10 weeks]
  The changes in deoxyhemoglobin driven by localized changes in brain blood flow and blood oxygenation associated with individual trial-by-trial reinforcement learning computational model parameters at the time of choice valuation (expected reward value during safe contexts and expected reward value during threat contexts) and choice outcome (reward prediction errors during safe contexts and reward prediction errors during threat contexts).

SECONDARY OUTCOMES:
Within-subject BOLD contrast for unexpected absence of juice vs. expected absence of juice (negative temporal Prediction Errors) for safe and threat contexts. | [10 weeks]
  The changes in deoxyhemoglobin driven by localized changes in brain blood flow and blood oxygenation between the unexpected absence of juice vs. expected absence of juice in safe contexts and threat contexts.
Within-subject BOLD contrast for the unexpected delivery of juice vs. the expected delivery of juice (positive temporal Prediction Errors) for safe and threat contexts. | [10 weeks]
  The changes in deoxyhemoglobin driven by localized changes in brain blood flow and blood oxygenation between the unexpected delivery of juice vs. the expected delivery of juice in both safe and threat contexts.
Within subject beta coefficients for each parametrically modulated regressor of an approach avoidance conflict task. | [10 weeks]
  The changes in deoxyhemoglobin driven by localized changes in brain blood flow and blood oxygenation associated with individual trial-by-trial reinforcement learning computational model parameters at the time of choice valuation (expected reward value, expected threat value, and conflict between reward and threat value), anticipation (expected reward and threat value), and choice outcome (reward and threat prediction errors).

OTHER OUTCOMES:
Change in total score of the Clinician Administered PTSD Scale for DSM-5 from baseline to 10 weeks | 10 weeks
  A structured clinical interview measure of PTSD symptom severity
Change in total score of the PTSD Checklist for DSM-5 from baseline to 10 weeks | 10 weeks
  A self-report measure of PTSD symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Fonzo, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- Health Discovery Building (HDB), 1601 Trinity St., Bldg B., Z0600, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No